CLINICAL TRIAL: NCT04203472
Title: Influence of Type of Inhaler on Cough Severity and Tolerance of Therapy in Patients With Cough Variant or Cough Predominant Asthma
Brief Title: Optimal Type of Inhaler in Cough Variant- or Cough Predominant Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marta Dąbrowska, Medical Researcher, Medical University of Warsaw
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Inhaler in CVA
Record Dates: First submitted 2019-09-02; First posted 2019-12-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Asthma; Cough Variant Asthma
Keywords: inhalation technique; Dry Powder Inhaler; pressurized Metered Dose Inhaler
MeSH Terms: conditions — Asthma; Cough-Variant Asthma

STUDY DESIGN:
Intervention Model Description: In all patients cough severity and tolerance of therapy will be analyzed during therapy with budesonide and/ or formoterol administered by DPI and MDI used in turn. Order of using different types of inhalers will be accidental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide or budeosonide/formoterol administered by DPI (Experimental): In every patient cough severity and tolerance of therapy will be analyzed during therapy with budesonide and/ or formoterol administered by DPI for 14 days
  Interventions: Device: Budesonid or budesonide/fomoterol administered by DPI
- Budesonide or budeosonide/formoterol administered by MDI (Active Comparator): In every patient inhaler will be changed and cough severity and tolerance of therapy will be analyzed during therapy with the same drugs administered by MDI . Order of using different types of inhalers will be accidental
  Interventions: Device: Budesonid or budesonide/fomoterol administered by MDI

INTERVENTIONS:
Device: Budesonid or budesonide/fomoterol administered by DPI — Miflonide Breezhaler 200 mcg or Oxodil Aerolizer 12 mcg
  Other Names: Miflonide or Miflonide and Oxodil
  Arms: Budesonide or budeosonide/formoterol administered by DPI
Device: Budesonid or budesonide/fomoterol administered by MDI — Budiair 200 mcg or Atimos 12 mcg
  Other Names: Budiair or Budiair and Atimos
  Arms: Budesonide or budeosonide/formoterol administered by MDI

SUMMARY:
Asthma management is based on inhaled therapy, mainly on inhaled glucocorticosteroids (ICS). The efficacy of inhaled therapy depends on type of inhaler and proper inhalation skills. Additionally, in cough variant- or cough predominant asthma aerosol or dry powder of inhaler may tease upper airway and induce cough.

The aim of the study is to analyze if type of inhaler (DPI vs MDI) affects the efficacy of the management in cough variant or cough predominant asthma.

Twenty two patients with cough variant- or cough predominant asthma will be enrolled into the study.

Initially cough severity (in VAS scale), cough related quality of life (in Leicester Cough Questionnaire, LCQ) and number of cough episodes during 2 hours will be estimated. Additionally Asthma Control Test (ACT), Asthma Quality of Life Questionnaire (AQLQ) and spirometry will be performed.

Then, budesonide or budesonide and formoterol will be used in Aerolizer / Breezhaler or pMDI in turn (each for 14 days) in the same doses. Inhalation technique will be checked and if needed corrected.

After 14 days and then after 28 days, cough severity, LCQ, number of cough episodes, ACT, AQLQ, spirometry and inhalation technique will be assessed.

The results will be based on differences in cough severity, cough related quality of life, asthma related quality of life, control of asthma and number of cough episodes between therapy with DPI and MDI.

DETAILED DESCRIPTION:
Cough may be caused by both cough variant asthma or cough predominant asthma in 20-30% adults with chronic cough. Asthma management is based on inhaled therapy, mainly on inhaled glucocorticosteroids (ICS). The efficacy of inhaled therapy depends on type of inhaler and proper inhalation skills (1-2). Many of patients with asthma (as well as with COPD) make mistakes during inhaling, what negatively affect efficacy of management (3-4). Additionally, in cough variant- or cough predominant asthma aerosol or dry powder of inhaler may tease upper airway and induce cough (5).

Therefore aim of the study is to analyze if type of inhaler (Dry Powder Inhaler, DPI vs pressurized Metered Dose Inhaler, MDI) affects the efficacy of the management in cough variant or cough predominant asthma.

In all patients cough severity and tolerance of therapy will be analyzed during therapy with budesonide and/ or formoterol administered by DPI and MDI used in turn. Order of using different types of inhalers will be accidental.

Twenty two patients with cough variant- or cough predominant asthma will be enrolled into the study.

The sample size for the study was determined assuming that initially cough severity is at least 50/100 mm in VAS scale and minimal difference will be 20/100 mm. Providing these conditions, the sample size is 18 patients (α error 5%, power 80%); the sample was increased by 20% assuming drop out during the study.

Initially cough severity (in 10 mm VAS scale), cough related quality of life (in Leicester Cough Questionnaire, LCQ) and number of cough episodes during 2 hours will be estimated. Additionally Asthma Control Test (ACT), Asthma Quality of Life Questionnaire (AQLQ) and spirometry will be performed.

Then, budesonide or budesonide and formoterol will be stared in Aerolizer / Breezhaler or pMDI. Inhalation technique will be checked and if needed -corrected.

After 14 days, cough severity, LCQ, number of cough episodes, ACT, AQLQ, spirometry and inhalation technique will be assessed.

Then, type of inhaler will be changed, but the same doses of ICS and LABA will be administered. Once again inhalation technique will be checked and corrected if needed.

After 28 days, cough severity, LCQ, number of cough episodes, ACT, AQLQ, spirometry and inhalation technique will be assessed again.

The results will be based on differences in cough severity, cough related quality of life, asthma related quality of life, control of asthma and number of cough episodes between therapy with DPI and MDI.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for participating in the study
* Age ≥18 years
* Cough variant asthma or cough predominant asthma diagnosed and treated with inhaled corticosteroids (ICS) regularly at least 8 weeks prior to enrollment

Exclusion Criteria:

* Lack of informed consent
* Age <18 years
* Diagnosis of cough variant- or cough predominant asthma shorter than 8 weeks before enrollment
* Symptoms of infection or asthma exacerbation 4 weeks prior to beginning of the study or during the study
* Comorbidity that could prevent patient from using DPI or MDI (i e. advanced vision disorders, some mental diseases, advanced neurological diseases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
change in cough severity | 14 days and 28 days
  Assessment by 10 mm Visual Analogue Scale
change in cough related Quality of Life | baseline ,14 and 28 days
  Assessment by cough related Leicester Quality of Life Questionnaire (LCQ)

SECONDARY OUTCOMES:
change in asthma control | baseline , 14 and 28 days
  Assessment by Asthma Control Test
change in asthma related Quality of Life | baseline ,14 and 28 days
  Assessment by Asthma Quality of Life Questionnaire (AQLQ)
change in number of cough episodes counted per 2 hours | baseline, 14 and 28 days
  measured by investigator during visit

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Result] Morice AH, McGarvey L, Pavord I; British Thoracic Society Cough Guideline Group. Recommendations for the management of cough in adults. Thorax. 2006 Sep;61 Suppl 1(Suppl 1):i1-24. doi: 10.1136/thx.2006.065144. No abstract available. PMID 16936230
- [Result] Irwin RS, Baumann MH, Bolser DC, Boulet LP, Braman SS, Brightling CE, Brown KK, Canning BJ, Chang AB, Dicpinigaitis PV, Eccles R, Glomb WB, Goldstein LB, Graham LM, Hargreave FE, Kvale PA, Lewis SZ, McCool FD, McCrory DC, Prakash UBS, Pratter MR, Rosen MJ, Schulman E, Shannon JJ, Hammond CS, Tarlo SM. Diagnosis and management of cough executive summary: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):1S-23S. doi: 10.1378/chest.129.1_suppl.1S. No abstract available. PMID 16428686
- [Result] Inhaler Error Steering Committee; Price D, Bosnic-Anticevich S, Briggs A, Chrystyn H, Rand C, Scheuch G, Bousquet J. Inhaler competence in asthma: common errors, barriers to use and recommended solutions. Respir Med. 2013 Jan;107(1):37-46. doi: 10.1016/j.rmed.2012.09.017. Epub 2012 Oct 23. PMID 23098685
- [Result] Price DB, Roman-Rodriguez M, McQueen RB, Bosnic-Anticevich S, Carter V, Gruffydd-Jones K, Haughney J, Henrichsen S, Hutton C, Infantino A, Lavorini F, Law LM, Lisspers K, Papi A, Ryan D, Stallberg B, van der Molen T, Chrystyn H. Inhaler Errors in the CRITIKAL Study: Type, Frequency, and Association with Asthma Outcomes. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):1071-1081.e9. doi: 10.1016/j.jaip.2017.01.004. Epub 2017 Mar 9. PMID 28286157
- [Result] Kamimura M, Izumi S, Hamamoto Y, Morita A, Toyota E, Kobayashi N, Kudo K. Superiority of nebulized corticosteroids over dry powder inhalers in certain patients with cough variant asthma or cough-predominant asthma. Allergol Int. 2012 Sep;61(3):411-7. doi: 10.2332/allergolint.11-OA-0357. Epub 2012 May 25. PMID 22627846